CLINICAL TRIAL: NCT03472339
Title: A Randomized Double-blinded Trial Comparing the Clinical Efficacy and Pharmacokinetic Parameters of Oral Diclofenac and Intramuscular Diclofenac in Patients With Acute Limb Injuries
Brief Title: Clinical Trial Comparing Intravenous and Oral Diclofenac and Pharmacokinetics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Isma Qureshi, Academic Research Associate, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16413/16
Record Dates: First submitted 2018-03-01; First posted 2018-03-21 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Pain Management; Limb Injury
Keywords: Acute limb injury, Diclofenac, pain management
MeSH Terms: conditions — Agnosia | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: Double blind randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: A computer generated block randomization sequence will be generated and stored with sequential coding known to the clinical pharmacist only. Within the randomization another stratified randomized sequence will be generated, for the patients to be enrolled for the PK study. Among the 300 trial packets prepared for the study, 20 packets will contain one additional code that will indicate the subject to be enrolled in the PK study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): diclofenac sodium75 mg, intravenously, once
  Interventions: Drug: Diclofenac Sodium
- Group B (Active Comparator): diclofenac sodium 100 mg, orally, once
  Interventions: Drug: Diclofenac Sodium

INTERVENTIONS:
Drug: Diclofenac Sodium — Group A-Intramuscular diclofenac sodium+oral placebo Group B-Oral diclofenac sodium+ intramuscular placebo

SUMMARY:
NSAIDs are commonly used in the management of acute pain; Diclofenac is one from the same class. It is an amino phenyl acetic acid derivative which inhibits prostaglandin biosynthesis to produce analgesic, antipyretic and anti-inflammatory effect. The drug efficacy and safety in acute pain management has been proved by several studies like in renal colic, post and pre-operative pain management, migraines etc. It's also known to have an opioid-sparing effect. Mode of administration is one of the important factors to consider in a busy emergency room. Perception about the route of administration differs among patients. As believed,injectable have rapid onset, easier to titrate, and patients respond better to them as they consider them stronger than oral medication. Number of trials has compared oral and parenteral NSAIDs. Most found no benefit to the parenteral route. Considering the limitations of the previously done studies like small sample size, heterogeneity in the group of patients enrolled, improper blinding and comparing of two different drugs from the same class. Therefore, aim of the study is to conduct a Double blind randomized clinical trial to assess the clinical efficacy and pharmacokinetic parameters of oral diclofenac compared to intramuscular diclofenac in patients with acute limb injury.

In this two group double blind randomized clinical trial, the clinical efficacy and pharmacokinetic parameters among the two groups will be assessed. Eligible patients visiting to HGH-ED, age (above 18 years) with acute limb injury, having moderate to severe pain (defined as pain score of >=4 on Numerical rating scale) will be recruited. With the use of computer generated block randomization, subjects will be allocated to one of the two treatment groups in the ratio of 1:1. Each group will receive either (intramuscular diclofenac / oral placebo) or (oral diclofenac / intramuscular placebo). Among the 300 subjects enrolled for the study, further stratified randomization will be done in order to enroll 20 patients for pharmacokinetic study within the subjects.High-performance liquid chromatography, method will be used for the determination of drug concentration in human plasma, for detailed pharmacokinetics. The pain score will be assessed by using the validated pain scale i.e. Numerical rating scale (NRS). The participants, clinicians and investigators will be masked to treatment assigned and the results will be analyzed by the intention to treat analysis among the two group treatment.

DETAILED DESCRIPTION:
This will be a prospective, double blinded, randomized clinical trial, and it will be conducted and reported according to the consolidated standards of reporting trials group 14.

Setting:

The study will be conducted at Hamad General Hospital Emergency Department (HGH-ED). Since it is the largest tertiary care medical center in the country, having a busy ED with monthly census exceeding 40,000 (approximately 500,000 annually). Patients with acute limb injury are frequently seen in ED.

Sample size calculation:

300 patients are required to have a 95% chance of detecting, as significant at the 5%level, a decrease in the primary outcome measure from 70% in the control group to 50% in the experimental group. As for the number of subjects to be enrolled in pharmacokinetic study is directly related to both power and cost of the trial (14)*, we aim a convenience sample of 20 subjects, 10 in each group.

Screening and Randomization:

All adult patients (age above 18-65 years) presenting with Acute limb injury will be assessed by the available physician initially. Patient's hospital identification number will be put into the study registry. The registry will assure all consecutive patients are screened. Once an eligible patient is identified the physicians will page the research assistant, who will be available in the emergency department from 6 am to 2 pm on week days. After meeting the inclusion criteria and the subject agrees to participate, written consent will be obtained. The enrolled participants will be randomly assigned in a 1:1 ratio, to one of the two groups- either intramuscular diclofenac or oral diclofenac, from the trial packet available in the stock.

A computer generated block randomization sequence will be generated and stored with sequential coding known to the clinical pharmacist only. Within the randomized sequence, another stratified randomized sequence will be generated for the 20 subjects to be enrolled for pharmacokinetic trial only during the morning shifts. In case of adverse reaction form will be filled and medical research center will be notified for such event.

Intervention:

Typical trial packet

* Syringe A: 3ml solution, diclofenac 75mg or placebo
* Tablet: 100mg diclofenac tablet or placebo A trial packet will contain one syringe labelled A (3ml) and one tablet labelled B (100mg) in an amber colored zip lock pouch. Each will be labelled with a sticker mentioning a unique code, date of preparation and instructions for administration.

Trial packs A B Combination 1 Intramuscular Diclofenac Oral Placebo Combination 2 Oral Diclofenac Intramuscular Placebo Trial packs will be prepared and kept in a locker ready to be used on a daily basis. The team preparing these packets will have no further part in patient treatment or data recording.

Dosage

* Intramuscular Diclofenac will be available in 75mg/3ml concentration for single dose intramuscular administration.
* Tablet Diclofenac will be available as 100mg tablet for single dose per oral administration.

The protocol dictates to administer syringe "A" (3ml) intramuscular, 100mg tablet labeled "B" to administer per oral.

Data and sample collection:

Patient enrolled for pharmacokinetic measurement, will have an intravenous line to obtain blood for routine sampling, a hep- lock will be attached to the line, for the withdrawal of repeated samples. Blood samples will be collected only in weekdays and morning shifts from 6am until 2 pm. 3 ml of blood will be withdrawn at time 0, 5, 10, 15, 20, 25, 30, 45 and 60 minutes. High- performance liquid chromatography method will be used to determine drug in human plasma as the method is potentially considered to be used for detailed pharmacokinetics, pharmacodynamics and bioequivalence studies of diclofenac in humans. Along with blood sampling patient pain score using a numerical rating scale (NRS) will be used to assess the pain, as for the rest of the patients. Pain scores will be recorded at 0, 5, 10, 15, 20, 25, 30, 45 and 60, minutes following administration of analgesia. Patients reported pain scores will be recorded contemporaneously and patient will not be reminded of the previous score. If patients pain does not reduce significantly at the end of 30 minutes after receiving the study drug, a rescue analgesia in the form of morphine will be given 3mg intravenously every 5 minutes until sedation side effects or pain drops to Numerical rating score = or <2.Patient will be discharged as per the advice of the available physician in ED.

ELIGIBILITY:
Eligible patients are those adults (age at least 18years), presenting to HGH-ED with complaints of acute limb injury, initially evaluated by the physician.

Inclusion criteria:

1. Healthy volunteers
2. Adult patients above 18-65 years of age.
3. Patients with soft tissue injury/ cut wounds
4. Pain score more than or equal to 4 on NRS.
5. Patients weight more than or equal to 50kgs.
6. If treating physician approves patient participation in the study.
7. Not on any medication.

Exclusion criteria:

1. Received any analgesic within last 12 hours, on the day of visit to ED.
2. Patients with fractures
3. Allergic to diclofenac.
4. Cardio-vascular disease, renal impairment, stroke or any other co-morbidity / chronic illness.
5. Pregnancy / Nursing
6. Peptic ulcers
7. Bleeding disorders
8. liver disease
9. Bronchial asthma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-04-15 (Estimated); Study Completion 2018-04-15 (Estimated)

PRIMARY OUTCOMES:
Difference in proportion of patients achieving 50% pain reduction | 30 mins
  The primary outcome is defined as the proportion of patients achieving pain reduction by 50% at 30 minutes following analgesia administration.
the mean difference in plasma concentration for two drugs | 60 mins
  Cmax - Peak plasma concentration and Time curve

SECONDARY OUTCOMES:
proportion of patients achieving pain reduction of >=2 Numerical Rating Scale( which is a numeric scale where respondent selects a whole number from 0 to 10, where 0 means no pain and 10 means worst pain) from the initial score | at 30 mins
  to assess proportion of patients who could achieve minimal significant pain reduction
Rescue analgesia | after 30 mins
  proportion of patients requiring a rescue analgesia after 30 min in each group
Adverse events | 2 hours
  the number of adverse events in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Isma Qureshi, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derry P, Derry S, Moore RA, McQuay HJ. Single dose oral diclofenac for acute postoperative pain in adults. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD004768. doi: 10.1002/14651858.CD004768.pub2. PMID 19370609
- [Background] Marret E, Kurdi O, Zufferey P, Bonnet F. Effects of nonsteroidal antiinflammatory drugs on patient-controlled analgesia morphine side effects: meta-analysis of randomized controlled trials. Anesthesiology. 2005 Jun;102(6):1249-60. doi: 10.1097/00000542-200506000-00027. PMID 15915040
- [Background] Pathan SA, Mitra B, Straney LD, Afzal MS, Anjum S, Shukla D, Morley K, Al Hilli SA, Al Rumaihi K, Thomas SH, Cameron PA. Delivering safe and effective analgesia for management of renal colic in the emergency department: a double-blind, multigroup, randomised controlled trial. Lancet. 2016 May 14;387(10032):1999-2007. doi: 10.1016/S0140-6736(16)00652-8. Epub 2016 Mar 16. PMID 26993881
- [Background] Gan TJ, Daniels SE, Singla N, Hamilton DA, Carr DB. A novel injectable formulation of diclofenac compared with intravenous ketorolac or placebo for acute moderate-to-severe pain after abdominal or pelvic surgery: a multicenter, double-blind, randomized, multiple-dose study. Anesth Analg. 2012 Nov;115(5):1212-20. doi: 10.1213/ANE.0b013e3182691bf9. Epub 2012 Aug 10. PMID 22886837
- [Background] Turturro MA, Paris PM, Seaberg DC. Intramuscular ketorolac versus oral ibuprofen in acute musculoskeletal pain. Ann Emerg Med. 1995 Aug;26(2):117-20. doi: 10.1016/s0196-0644(95)70138-9. PMID 7618770
- [Background] Ucar R, Biyik M, Ucar E, Polat I, Cifci S, Ataseven H, Demir A. Rectal or intramuscular diclofenac reduces the incidence of pancreatitis afterendoscopic retrograde cholangiopancreatography. Turk J Med Sci. 2016 Jun 23;46(4):1059-63. doi: 10.3906/sag-1502-104. PMID 27513404